CLINICAL TRIAL: NCT03734601
Title: Very Low-dose Total Body Irradiation in Combination With Total Lymphoid Irradiation and Anti-Thymocyte Globulin to Improve Donor Engraftment in Patients Undergoing Non-Myeloablative Hematopoietic Cell Transplantation
Brief Title: Total Body Irradiation +/- Total Lymphoid Irradiation & Anti-Thymocyte Globulin in Non-myeloablative Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Lowsky, Professor of Medicine (Blood and Marrow Transplantation and Cellular Therapy), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-47407; BMT330 (Other: OnCore ID); IRB-47407 (Other: Stanford IRB)
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorder; Chronic Lymphocytic Leukemia; B-cell Lymphoma; T-cell Lymphoma; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myelomonocytic, Chronic | interventions — Whole-Body Irradiation; Antilymphocyte Serum; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBI+TLI (Experimental): TBI, single exposure on Day -1, 80 centigray (cGy) in addition to total lymphoid irradiation (TLI, 120 cGy/day for 9 days, weekends excluded) and anti-thymocyte globulin (ATG) 1.5 mg/kg (conditioning regimen)
  Interventions: Radiation: Total body irradiation (TBI); Drug: Anti-thymocyte globulin (ATG); Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF); Radiation: Total lymphoid irradiation (TLI)

INTERVENTIONS:
Radiation: Total body irradiation (TBI) — Administer Total body irradiation (TBI) 80 cGy on Day 1 of standard TLI ATG conditioning
Drug: Anti-thymocyte globulin (ATG) — Given intravenous (IV), Dose 1.5 mg/kg x 5 days
Drug: Tacrolimus — Oral, Dose 0.05 mg/kg twice daily, can be given intravenous (IV)
  Other Names: Fujimycin
Drug: Mycophenolate mofetil (MMF) — Given Oral, 15 mg/k every 2 hours for peripheral blood stem cells (PBSC) from matched related donors; 15 mg/kg every 8 hours for PBSC from unrelated donors (URDs) or mismatched related donors.
  Other Names: Cellcept; MMF
Radiation: Total lymphoid irradiation (TLI) — 9 x 120 cGy over 11 days

SUMMARY:
The purpose of this study is to evaluate whether addition of a low dose of total body irradiation (TBI) to a standard preparation for transplant [total lymphoid irradiation (TLI) and anti-thymocyte globulin (ATG)] conditioning will help to augment donor chimerism without reducing tolerability of this regimen or increasing the risk of graft-vs-host disease (GVHD)

DETAILED DESCRIPTION:
Primary Objective:

• Determine the proportion of patients with full donor T-cell chimerism at Day 28 following hematopoietic cell transplantation.

Secondary Objectives:

* Determine the risk of disease progression, overall and event free survival, and non-relapse mortality, following treatment with TLI; ATG; and TBI.
* Determine the incidence of acute and chronic GVHD following treatment with TLI; ATG; and TBI.

Exploratory Objectives:

• Determine the changes in frequency of hematopoietic stem, progenitor, and mature cell subsets and the changes in cytokine milieu and cellular architecture in the bone marrow of patients receiving TLI compared to TLI+TBI.

ELIGIBILITY:
INCLUSION CRITERIA

* Has a human leukocyte antigen (HLA)-matched or single allele mismatched adult sibling donor or unrelated donor.
* Acute myeloid leukemia (AML); myelodysplastic syndrome (MDS); myeloproliferative disease syndrome (MPD)]; chronic lymphocytic leukemia (CLL); B- or T-cell non Hodgkin lymphoma (NHL); Hodgkin lymphoma (HL); or chronic myelomonocytic leukemia (CMML), suitable for treatment with allogeneic transplant after TLI and ATG reduced intensity conditioning.
* Considered at high-risk for regimen-related toxicity from fully-ablative transplant conditioning (therefore reduced-intensity conditioning is recommended).
* Ability to understand and the willingness to sign a written informed consent document. Patients must have signed informed consent to participate in the trial.

EXCLUSION CRITERIA

* Uncontrolled bacterial, viral or fungal infection defined as currently taking medication and progression of clinical symptoms.
* Progressive hemato lymphoid malignancy despite conventional therapy.
* Chronic myelogenous leukemia (CML).
* Active CNS involvement of the underlying malignancy.
* HIV positive
* Pregnant or lactating
* Prior malignancy (EXCEPTION: diagnosed > 5 years ago without evidence of disease, OR treated ≤ 5 years ago but have a greater than 50% chance of life expectancy of ≥ 5 years for that malignancy).
* Have a psychiatric disorder(s) or psychosocial circumstance(s) which in the opinion of the primary physician would place the patient at an unacceptable risk from transplant.
* Left ventricular ejection fraction (LEVF) < 30%, or uncontrolled cardiac failure
* Diffusing capacity of lung for carbon monoxide (DLCO) < 40% predicted
* Total bilirubin > 3 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) > 4 x upper limit of normal (ULN)
* Creatinine > 2 mg/dL and an estimated creatinine clearance < 40 mL/min
* Poorly-controlled hypertension despite multiple antihypertensive medications
* Karnofsky Performance Status (KPS) < 60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TBI+TLI
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Full-dose Donor Chimerism (FDC) at Day 28 Following TLI/ATG/TBI Conditioning.
Description: Subsequent to TLI/ATG/TBI conditioning, the proportion of participants with full dose donor chimerism (FDC) will be determined by Day 28. FDC is defined as achieving ≥ 95% donor type in the CD3+ lineage within 28 days of donor cell infusion, as assessed by short tandem repeat (STR) testing. The outcome will be expressed as the number of participants that achieve FDC by Day 28, a number without dispersion.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants | 13

2. Secondary Outcome: Disease Progression
Description: Transplant recipients will be assessed for disease progression at 1 year after hematopoietic cell transplantation (HCT). The outcome is reported as the number of transplant recipients who experienced disease progression.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants | 7

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the number of transplant recipients remaining alive at 12 months after transplant. The outcome is expressed as the number of transplant recipients who remained alive at 12 months after treatment, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants | 16

4. Secondary Outcome: Event-free Survival (EFS) at 1 Year
Description: Event-free survival (EFS) is defined as the number of transplant recipients remaining alive at 12 months after transplant and who did not experience disease relapse defined as blasts < 5%. The outcome is expressed as the number of transplant recipients remaining alive at 12 months after transplant without disease relapse, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants | 16

5. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Non-relapse mortality (NRM) is defined as death without known disease relapse or recurrence. The outcome is expressed as the number of transplant recipients whose cause of death was not disease relapse or recurrence, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants | 2

6. Secondary Outcome: Graft vs Host Disease (GvHD)
Description: Recipients will be monitored for Grade 2 to 4 graft vs host disease (GvHD). The outcome is reported as the number of transplant recipients who experienced acute GvHD grades 2 to 4, the number of transplant recipients who experienced chronic and extensive GvHD. In addition, the number of transplant recipients with chronic and extensive GvHD that was refractory to treatment ("persistent") is reported. Per protocol, the result for chronic extensive and persistent GvHD is based on the subset of participants that had chronic and extensive GvHD.
Time Frame: 1 year
Population: Per protocol, the outcome for chronic extensive and persistent GvHD is based on the subset of participants that had chronic and extensive GvHD.
Measure: Count of Participants; unit: Participants
Arm/Group | TBI+TLI
Number analyzed (Participants) | 22
Participants
  Acute GvHD | 5
  Chronic extensive GvHD | 8
  Chronic extensive and persistent GvHD: number analyzed (Participants) | 8
  Chronic extensive and persistent GvHD | 3

ADVERSE EVENTS:
Time Frame: 60 days, except collection of mortality information was open-ended.
Description: Per protocol, adverse event collection was limited, as follows.
  * Non-serious adverse event collection was limited to Grade 1 to 3 events that resulted in participant termination or withdrawal from the study
  * Serious adverse events, and details of, were only collected for 60 days after the transplant.
  * Mortality collection was open-ended.
Arm/Group | TBI+TLI
All-Cause Mortality (participants affected / at risk) | 6/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI+TLI (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Chronic graft vs host disease (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03734601/Prot_SAP_001.pdf